CLINICAL TRIAL: NCT06745947
Title: Development of a Behavioral Economic Intervention to Improve HIV-related Behaviors Among Sexual Minority Individuals
Brief Title: Behavioral Economic Intervention to Improve HIV Behaviors in Sexual Minority Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Chukwuemeka Okafor, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000869; R34DA060078 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: HIV Prevention
Keywords: HIV negative; Methamphetamine use; HIV PrEP medication

STUDY DESIGN:
Intervention Model Description: A two-arm pilot randomized controlled trial
Who Masked: Investigator
Masking Description: Although it is not possible to fully blind participants due to the nature of the EFT intervention, research staff responsible for outcome assessments (e.g., PrEP adherence, methamphetamine use, and sexual risk behaviors) will be blinded to the participants' group assignment to minimize assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Episodic Future Thinking App (Experimental): EFT is a behavioral economic intervention designed to improve decision-making by reducing delay discounting and improving demand. The EFT intervention will be administered through a combination of in-person counseling sessions and mobile health (mHealth) technology via an app platform.
  Interventions: Behavioral: EFT
- Control Group (No Intervention): Standard of Care: The standard of care group will receive brief information and supportive counseling around PrEP adherence, methamphetamine use reduction and engaging in safe sexual behaviors. Participants will also receive counseling on a topic of concern identified by the participant.

INTERVENTIONS:
Behavioral: EFT — Participants who meet the eligibility criteria will receive the EFT intervention, a cognitive training exercise designed to help them generate and visualize future events or goals. The intervention will be administered individually, in person, by a trained counselor
  Other Names: Episodic Future Thinking
  Arms: Episodic Future Thinking App

SUMMARY:
This research study is testing a new behavioral therapy called Episodic Future Thinking or EFT can help people reduce drug use and risky sexual behaviors while helping them adhere to their HIV prevention medication (PrEP). Participants will be randomly assigned to one of two groups. One group will receive standard care, which includes counseling on HIV prevention, drug use reduction, and sexual health. The other group will receive standard care plus a new program called Episodic Future Thinking (EFT), where participants will think about and plan for their future goals using a mobile app and counseling sessions. Study procedures that are not part of regular care include filling out surveys, providing blood, urine, and swab samples for testing, and using the EFT app.

DETAILED DESCRIPTION:
Phase 1 of the study will involve a formative evaluation of the Episodic Future Thinking (EFT) intervention among (n=10) sexual minority individuals (SMIs) utilizing qualitative interviews. (This phase of the study data will not be reported on ClinicalTrials.gov, since it is not part of the randomized controlled trial).

Phase 2 of the study will utilize a two-arm pilot randomized controlled trial of Episodic Future Thinking plus standard of care (intervention) vs. standard of care only (control) condition to improved HIV-related behaviors (PrEP adherence, sexual risk behaviors and methamphetamine use) among sexual minority individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 - 34 years of age
* HIV negative (assessed via Rapid HIV Antibody Test)
* Identify as gay, or bisexual
* Recent (past 3 months) methamphetamine use
* Currently prescribed and taking HIV PrEP medication
* Self-reported HIV PrEP nonadherence in the past three months
* Urine screen test for PrEP nonadherence
* Self-reported condomless anal sex or a STI in the past three months
* Able to attend all study visits
* Fluent in English

Exclusion Criteria:

* Currently receiving treatment for any substance use disorder,
* HIV positive
* Having a medical or psychiatric illness that in the opinion of the PI would interfere with study participation
* Unable to provide informed consent
* Unable to attend protocol directed study visits
* Any plans that would preclude study completion (e.g. surgery, major medical treatments such as chemotherapy, incarceration, travel/moving out of San Antonio, Texas)

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The proposed research will specifically target sexual minority individuals (SMI) for recruitment including individuals who are cisgender and transgender.
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Dried Blood Spot Analysis for PrEP adherence | Day 1 to Day 180
  Blood spots will be collected and assessed for PrEP adherence. Number of subjects adhering to PrEP will be reported.
Urine Collection for Drug Screening | Day 1 to Day 180
  Urine will be tested for drug screening. Number of subjects that result in a negative drug screening will be reported.
Urine Collection for Sexually Transmitted Infections (STIs) | Day 1 to Day 180
  Urine will be tested for STIs. Number of subjects that test negative for STIs will be reported.
Rectal Swab for STI testing | Day 1 to Day 180
  A rectal swab will be obtained for STI. Number of subjects that test negative for STIs will be reported.
Pre-exposure Prophylaxis (PrEP) Related Intentions | Day 1 to Day 180
  A 3-item scale to measure PrEP-related intentions (e.g., "During the next three months, I will talk to a health care provider about PrEP"; "During the next three months, I will seek out more information about PrEP" and "During the next three months, I will get a prescription for PrEP"). Response options will be 1 = No, definitely not; 2 = No, probably not; 3 = Yes, probably and 4=Yes, definitely. A total range of scores is 3-12 with a higher score indication a greater intention of taking preventative measures.
PrEP Attitudes | Day 1 to Day 180
  A 5-item scale to evaluate attitudes regarding PrEP use (e.g., "People who take PrEP are responsible"; "Taking PrEP is safe"). Response options will range from 1=strongly disagree to 5=strongly agree. Total scores will range between 5 and 25, with higher scores indicating more favorable attitudes toward PrEP use.
PrEP Stigma | Day 1 to Day 180
  A 5-item scale to assess PrEP stigma (e.g., "People who take PrEP are promiscuous"). Responses will be on a 5-point scale, ranging from 1=strongly disagree to 5=strongly disagree. The total range of scores is 5-25, where higher scores denote greater stigma associated with PrEP.
PrEP Self-efficacy | Day 1 to Day 180
  Participants will self-report the level of difficulty they anticipate in performing 8 behaviors associated with PrEP use (e.g., "How difficult would it be for you to seek out more information about PrEP to decide if it is right for you?"). Responses will be on a scale from 1=very hard to do to 4=very easy to do. Total scores range from 8-32, where higher scores suggest higher levels of self-efficacy.

SECONDARY OUTCOMES:
Rapid HIV test | Day 30 to Day 180
  Test for HIV infection. Number of negative results will be reported.
Delayed Discounting | Day 1 to Day 180
  Delay discounting tasks will consist of 1) a standard adjusting-amount monetary tasks presenting repeated choices between various amounts of money now ($0 to $1,000) and $1,000 after a fixed delay (1 day to 25 years); 2) a cross-commodity task presenting choices between various amounts of methamphetamine now and money later in which the values are made equivalent with the monetary task; and 3) a condom delay discounting task assessing the likelihood that the participant would have sex with their ideal partner immediately with no condom vs. with a condom following a delay. Delayed discounting rate (or k) is an index of the devaluation of a rewards over time, with higher k values representing steeper discounting rates and a greater preferences for immediate rewards.
Demand | Day 1 to Day 180
  Demand tasks will consist of hypothetical purchasing tasks assessing 1) Methamphetamine demand (grams of methamphetamine purchased as a function of increasing price); 2) condom demand (likelihood of purchasing condoms as a function of increasing price, with the follow-up question of whether they do not have sex or have sex without a condom when the likelihood of condom purchasing goes to zero); and 3) PrEP demand (likelihood of purchasing a one-month supply of PrEP as a function of increasing price). Demand data will be fit to an exponentiated demand model: Q=Q0*10k(e-αQ0C-1), where Q represents consumption/use of the commodity as a function of increasing cost (C).
Diagnostic and Statistical Manual of Mental Disorders (DSM)-5-TR Self-rated Level 1 | Day 1 to Day 180
  This adult version of the measure consists of 23 questions that assess 13 psychiatric domains, including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. Each item inquires about how much (or how often) the individual has been bothered by the specific symptom during the past 2 weeks. Each item on the measure is rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day).
  Scoring:
  Scoring can be done at three levels:
  Item Level: Review individual item scores. Domain Level: Sum item scores within each domain. Full Survey Level: Sum all item scores.
Generalized Anxiety Disorder Screener (GAD-7) | Day 1 to Day 180
  The GAD-7 will be used to assess generalized anxiety symptomology. This is a 7-item measure that asks participants to rate the frequency with which they have been bothered by anxiety symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores on all items are summed up to obtain a total severity score between 0 and 28. Scores reflect no significant anxiety symptoms (0-4), mild anxiety symptoms (5-9), moderate anxiety symptoms (10-14), and severe anxiety symptoms (>15)

CONTACTS AND LOCATIONS:
Overall Officials: Emeka Okafor, PhD, MPH, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication policy will focus on ensuring that all dissemination of research findings from this study is conducted in an accurate, transparent and ethical manner. Authorship will be determined based on significant contributions to the study's conception, design, data acquisition, analysis or interpretation as well as in drafting and critically revising the manuscript. During this review process any potentially identifiable information will be carefully reviewed and anonymized if necessary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Summary results will be published through ClinicalTrials.gov and the study results will be published in a peer review journal after study completion and data analysis.